CLINICAL TRIAL: NCT05416892
Title: What is the Impact of Implementing Pharmaceutical Algorithms in the PharmaClass® Software, on the Handling the Patient's Medication Load, by the Clinical Pharmacist? Analysis of These Impacts Within 2 Geriatric Units of the CHU Brugmann Hospital
Brief Title: What is the Impact of Implementing Pharmaceutical Algorithms in the PharmaClass® Software, on the Handling the Patient's Medication Load, by the Clinical Pharmacist?
Status: Completed | Type: Observational
Sponsor: Murielle Surquin (Other)
Responsible Party: Sponsor-Investigator, Murielle Surquin, Head of Geriatry Department, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-PharmaClass
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Pharmacist-Patient Relations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients of Geriatric Wards SU06 and SU13 of the CHU Brugmann Hospital
  Interventions: Other: Pharmaclass® software

INTERVENTIONS:
Other: Pharmaclass® software — Clinical decision support tool via artificial intelligence in order to improve the patient's medication management.

SUMMARY:
The clinical pharmacists present in the hospitalisation units aim to ensure the daily review of the drug prescriptions of hospitalized patients.

In order to optimize their work, the objective of this study would be to provide them with a clinical decision support tool via artificial intelligence in order to improve the patient's medication management. This study will test the Pharmaclass® software.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patient entering the SU06 or SU13 geriatrics unit of the Paul Brien site of the CHU Brugmann Hospital between November 16 2021 and April 15, 2022
* Speaking French and/or Dutch
* With chronic renal failure or taking at least one medicine for diabetes, heart, COPD, asthma, high blood pressure, epilepsy, atrial fibrillation, osteoporosis, high cholesterol, pain, parkinsonism, blood clotting, constipation, thyroid, depression, benign prostatic hypertrophy, gastric ulcer, Alzheimer's disease, cirrhosis as well as for electrolyte disorders (hypo or hypernatremia / potassium / calcium/magnesemia/phosphatemia).

Exclusion Criteria:

* Patient who died or was transferred to another care unit during his/her hospitalization

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Hospitalized patient entering the SU06 or SU13 geriatrics unit of the Paul Brien site of the CHU Brugmann Hospital between November 16 2021 and April 15, 2022
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Time | 5 months
  Time required to perform an intervention (pharmacist versus software)
Dosage compliance | 5 months
  Dosage compliance with existing recommendations and laboratory results/clinical parameters (pharmacist versus software)
Medication error severity | 5 months
  Severity of the medication error that could be avoided (pharmacist versus software)
Geriatrician approval | 5 months
  Number of interventions validated/refused by the geriatrician (pharmacist versus software)

CONTACTS AND LOCATIONS:
Overall Officials: Charline DANNEEL, Principal Investigator — CHU Brugmann
Locations (1):
- Brugmann university hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No